CLINICAL TRIAL: NCT01130675
Title: Does Coffee Consumption Prevent or Shorten Postoperative Ileus After Colon Resection? A Prospective Randomized Clinical Trial
Brief Title: Does Coffee Consumption Prevent or Shorten Postoperative Ileus After Colon Resection?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-13493
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eight ounces of caffeinated coffee for breakfast and lunch (Active Comparator)
  Interventions: Other: caffeinated coffee
- standard care (No Intervention)

INTERVENTIONS:
Other: caffeinated coffee — 8 oz. of caffeinated cofee/breakfast&noon meal. No intervention for 2nd arm.
  Arms: eight ounces of caffeinated coffee for breakfast and lunch

SUMMARY:
The purpose of this study is to determine if consuming an 8 ounce cup of coffee with breakfast and lunch is effective in preventing or reducing postoperative ileus.

DETAILED DESCRIPTION:
Recent evidence has shown that a multimodal rehabilitation program can accelerate recovery of GI function after colon resection. 8 A multicenter, randomized, placebo-controlled, double-blind, phase 3 trial demonstrated that Alvimopan, a peripherally acting mu-opioid receptor antagonist, appears to accelerate GI tract recovery by 1 day, and reduces postoperative ileus-related morbidity without compromising opioid analgesia. 9 Asao et al demonstrated that gum chewing can accelerate recovery of GI function, also by 1 day, after abdominal surgery. 10 Epidural anesthesia has been shown to shorten duration of POI, as well as improve pain control, decrease pulmonary complications, and quicken recovery times. However, it does not appear to reduce overall length of stay. 4 However, Neudecker et al. were unable to reproduce the results of previous trials evaluating the effect of thoracic epidural analgesia on duration of postoperative ileus following laparoscopic sigmoid resection. 11 Given conflicting data, no one single measure has been adopted for the prevention POI.

Recent evidence has shown that coffee may be a stimulant for the GI Tract. A small study of 16 healthy volunteers demonstrated that coffee appears to increase rectal tone thus implying an impact on defecation mechanics.12 Furthermore, several studies have demonstrated caffeinated coffee to be a stimulant of motor activity in the colon.13,14 Given its potential pro-motility properties in the GI tract, it seems reasonable to postulate that coffee, a commonly consumed product by the general public, may play a role in shortening and possibly preventing POI. This directly impacts overall patient satisfaction but will reduce length of stay and overall hospital costs.

ELIGIBILITY:
Inclusion Criteria:

* Elective partial bowel resection with primary anastomosis for either cancer or benign disease.
* Laparoscopy or laparotomy

Exclusion Criteria:

* Total colectomy
* Colostomy
* Ileostomy
* Reversal of a stoma or synchronous resection
* Complete small or large bowel obstruction
* Scheduled to receive other treatments or techniques to reduce ileus

  1. epidural anesthetic tecniques
* Nasogastric tube for any length of timein the post-op period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Resolution of ileus | a mean difference of 24 hours to be significant
  Measured by hours to first flatus or bowel movement and tolerance of solid food.

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Memorial Medical Center Memorial Campus, Worcester, Massachusetts, United States